CLINICAL TRIAL: NCT04932382
Title: Misoprostol Prior to Intrauterine Device Insertion in Non-menstruating Women
Brief Title: Misoprostol Prior to Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MISO-IUD
Record Dates: First submitted 2021-06-12; First posted 2021-06-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: IUD
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol group (Other): 400 µg misoprostol vaginally ; these tablets will be introduced by the principal investigator, digitally without using speculum, 3 hours before IUD insertion into the posterior vaginal fornix of the woman while lying in the lithotomy position
  Interventions: Drug: Misoprostol; Device: IUD
- No misoprostol group (Other): will not receive any pre-insertion medications.
  Interventions: Device: IUD

INTERVENTIONS:
Drug: Misoprostol — will be used 3 h before IUD insertion
  Arms: Misoprostol group
Device: IUD — a copper T380A IUD

SUMMARY:
The intrauterine device (IUD) is a reliable, safe, long acting, and effective contraceptive method . In spite of that, the pain associated with IUD insertion can be a cause against its insertion. Many researches have been conducted aiming to decrease the degree of pain during IUD insertion; these studies included medical and also technical methods.

The physicians usually prefer to insert the IUD during women's menses because the women are very unlikely to be pregnant and the insertion is easier and the pain is lower The easiness of IUD insertion is a very important issue that can increase women's satisfaction and decrease insertion pain.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years
* Non-pregnant women
* Women who will come when there are non-menstruating.

Exclusion Criteria:

* Women received any analgesics or misoprostol in the 24 hours prior to insertion
* Women with any contraindications for IUD insertion
* Nulliparous women
* Women refuse to participate.
* Women have any contraindication of misoprostol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The degree of pain perception during IUD insertion assessed by visual analogue scale | 5 minutes
  The visual analogue scale scored from 0 to 10 degree, 0 degree means no pain while 10 degree means maximum pain

SECONDARY OUTCOMES:
The ease of IUD insertion: will be measured by visual analogue like scale [from 0 to 10] | 5 minutes
  0 means very easy insertion and 10 means so difficult insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided